CLINICAL TRIAL: NCT01617005
Title: Non-interventional Local Study to Describe the Safety, Tolerability and Efficacy of Tocilizumab in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-biologic DMARD
Brief Title: A Study of Tocilizumab in Participants With Active Rheumatoid Arthritis (RA) and an Inadequate Response to Non-Biological Disease-modifying Anti-rheumatic Drugs (DMARDs)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25699
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tocilizumab in Moderate to Severe Active RA: Moderate to severe active RA participants, receiving tocilizumab treatment according to effective official Summary of Product Characteristics (SPC), will be observed. The choice of therapy will be based exclusively on the medical decision of the treating physician before study enrollment. The study protocol does not enforce treatment initiation and also does not specify any treatment regimen.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive tocilizumab treatment according to effective official SPC. The study protocol does not enforce treatment initiation and also does not specify any treatment regimen.
  Other Names: RoActemra; L04AC07

SUMMARY:
This observational study will evaluate the safety and efficacy of tocilizumab in participants with active moderate to severe RA and an inadequate response to non-biologic DMARDs. Data will be collected from each eligible participant initiating tocilizumab treatment over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active RA (European League Against Rheumatism [EULAR] criteria)
* Inadequate response to DMARDs or tumor necrosis factor (TNF) antagonists
* Initiating treatment with tocilizumab according to SPC

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* Prior history or current inflammatory joint disease other than RA
* Previous treatment with any biological drug used in the treatment of RA
* Previous treatment with tocilizumab
* Any contraindication to treatment with tocilizumab
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following enrollment
* Pregnant women or nursing (breastfeeding) mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RA and an inadequate response to non-biologic DMARDs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Podgorica, Montenegro

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab in Moderate to Severe Active RA: Moderate to severe active Rheumatoid Arthritis (RA) participants, receiving tocilizumab treatment according to effective official Summary of Product Characteristics (SPC), were observed. The choice of therapy was based exclusively on the medical decision of the treating physician before study enrollment. The study protocol did not enforce treatment initiation and also did not specify any treatment regimen.
Period: Overall Study
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Started | 50
Completed | 48
Not Completed | 2
Not completed — Pregnancy | 1
Not completed — Lack of motivation for treatment | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- Tocilizumab in Moderate to Severe Active RA: Moderate to severe active RA participants, receiving tocilizumab treatment according to effective official SPC, were observed. The choice of therapy was based exclusively on the medical decision of the treating physician before study enrollment. The study protocol did not enforce treatment initiation and also did not specify any treatment regimen.
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs include both SAEs as well as non-serious AEs.
Time Frame: Baseline up to Week 24
Population: All participants enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Number analyzed (Participants) | 50
participants
  SAEs | 0
  AEs | 38

2. Secondary Outcome: Number of Participants With Good or Moderate Response According to European League Against Rheumatism (EULAR) Criteria
Description: EULAR response was based on 28-joint disease activity score (DAS28). The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline (CFB) in DAS28 score and the level of disease activity reached (absolute DAS28 score). Good responders had a CFB greater than (>) 1.2 with a DAS28 score less than or equal to (<=) 3.2; moderate responders had a CFB >1.2 with a DAS28 score >3.2 to <= 5.1 or a change from baseline >0.6 to <= 1.2 with a DAS28 score <= 5.1; non-responders had a CFB <=0.6 or CFB >0.6 to <=1.2 with DAS28 >5.1. Number of participants who achieved EULAR good response and EULAR moderate response were reported.
Time Frame: Baseline, Week 24
Population: All participants enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Number analyzed (Participants) | 50
participants
  EULAR Good Response | 0
  EULAR Moderate Response | 40

3. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to Lack of Efficacy
Time Frame: Baseline up to Week 24
Population: All participants enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Number analyzed (Participants) | 50
participants | 0

4. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Time Frame: Baseline up to Week 24
Population: As none of the participants discontinued treatment due to lack of efficacy, this outcome measure was not estimable.
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Arm/Group | Tocilizumab in Moderate to Severe Active RA
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 38/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab in Moderate to Severe Active RA (N=50)
Hypertension (Vascular disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 15
Leukopenia with neutropenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Gastralgia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hepatic transaminases increased (Investigations) | 10
Oral herpes simplex (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Fever (Infections and infestations) | 1
Bradycardia (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Polyartralgia (Musculoskeletal and connective tissue disorders) | 1
Hypercholesterolemia with hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.